CLINICAL TRIAL: NCT04315636
Title: Surfactant Nebulization for the Early Aeration of the Preterm Lung: a Single Blinded, Parallel, Randomized Controlled Trial
Brief Title: Surfactant Nebulization for the Early Aeration of the Preterm Lung
Acronym: SUNSET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sunset
Record Dates: First submitted 2020-03-06; First posted 2020-03-19 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Preterm Birth; Respiratory Distress Syndrome; Surfactant Deficiency Syndrome Neonatal
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surfactant nebulisation (Experimental): The experimental group will receive a positive end-expiratory pressure (PEEP, +/- noninvasive positive pressure ventilation) and nebulised surfactant via a customised vibrating membrane nebuliser. Nebulisation will commence with the first application of a PEEP and will continue for a maximum of 30 minutes.
  Interventions: Drug: Surfactant nebulisation
- Standard care (No Intervention): The control group will receive standard care (PEEP, +/- noninvasive positive pressure ventilation, without surfactant nebulisation).

INTERVENTIONS:
Drug: Surfactant nebulisation — 200 mg/kg body weight nebulised surfactant (Poractant alfa, Chiesi Farmaceutici SpA, Parma, Italy) via a customised vibrating membrane nebuliser (eFlow neonatal nebuliser system, PARI Pharma, Starnberg).
  Arms: Surfactant nebulisation

SUMMARY:
Respiratory distress syndrome is the most common cause of respiratory failure in preterm infants. Treatment consists of respiratory support and exogenous surfactant administration. Commonly, surfactant is administered via an endotracheal tube during mechanical ventilation. However, mechanical ventilation is considered an important risk factor for developing bronchopulmonary dysplasia.

Surfactant nebulisation during noninvasive ventilation may offer an alternative method for surfactant administration and has been shown to be promising in terms of physiological as well as clinical changes. In preterm infants with respiratory distress syndrome, the effect of intratracheally administered surfactant on lung function during invasive ventilation has been studied extensively. However, the effect of early postnatal surfactant nebulization remains unclear.

Therefore, the investigators plan to conduct a randomized controlled trial in order to investigate the effect of surfactant nebulization immediately after birth on early postnatal lung volume and short-term respiratory stability.

ELIGIBILITY:
Inclusion Criteria:

* inborn
* gestational age at birth from 26 0/7 to 31 6/7 weeks
* written informed consent

Exclusion Criteria:

* severe congenital malformation adversely affecting surfactant nebulisation or life expectancy
* a priori palliative care
* genetically defined syndrome

Max Age: 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
EIT: End-expiratory lung impedance (EELI) | Between birth and 30 minutes of life.
  Change in EELI using electrical impedance tomography (arbitrary units per kilogram)

SECONDARY OUTCOMES:
EIT: End-expiratory lung impedance (EELI) | At 6, 12, and 24 hours of life and at 36 weeks postmenstrual age
  EELI using electrical impedance tomography (arbitrary units per kilogram).
EIT: Regional ventilation distribution | At 6, 12, and 24 hours of life and at 36 weeks postmenstrual age.
  Regional ventilation distribution using electrical impedance tomography (arbitrary units per kilogram).
EIT: Tidal volumes | At 6, 12, and 24 hours of life and at 36 weeks postmenstrual age.
  Tidal volumes using electrical impedance tomography (arbitrary units per kilogram).
EIT: Association between EELI losses and SpO2/FiO2 ratio. | At 6, 12, and 24 hours of life.
  Association between the number of EELI losses >50% and the SpO2/FiO2 ratio.
EIT: Association between EELI losses and need/level of respiratory support. | At 6, 12, and 24 hours of life.
  Association between the number of EELI losses >50% and the need/level of respiratory support.
Physiological: Heart rate | For the first 30 minutes after birth, as well as at 6, 12, and 24 hours of life.
  Continuous recording of heart rate (beats per minute).
Physiological: Oxygen saturation (SpO2) | For the first 30 minutes after birth, and at 6, 12, and 24 hours of life.
  Continuous recording of SpO2 (%).
Physiological: Fraction of inspired oxygen | For the first 30 minutes after birth, and at 6, 12, and 24 hours of life.
  Continuous recording of fraction of inspired oxygen.
Physiological: SpO2/FiO2 ratio | At 6, 12, and 24 hours of life.
  SpO2/FiO2 ratio.
Physiological: Body temperature | In the delivery room.
  Number of events with body temperature <36.5 or >37.5°C.
Respiratory: Peak inspiratory pressure (PIP) | During the first 30 minutes of life.
  Continuous recording of PIP in the control group (cmH2O).
Respiratory: Positive end-expiratory pressure (PEEP) | During the first 30 minutes of life.
  Continuous recording of PEEP in the control group (cmH2O).
Respiratory: Tidal volume (Vt) | During the first 30 minutes of life.
  Continuous recording of Vt in the control group (cmH2O).
Respiratory: PEEP (positive end-expiratory pressure) | At 6, 12, and 24 hours of life.
  PEEP during noninvasive and invasive ventilation [mbar]
Respiratory: PIP (peak inspiratory pressure) | At 6, 12, and 24 hours of life.
  PIP during noninvasive and invasive ventilation [mbar]
Respiratory: Respiratory rate | At 6, 12, and 24 hours of life.
  Respiratory rate during noninvasive and invasive ventilation [breaths per minute]
Clinical: Length and type of noninvasive respiratory support | During the first 30 minutes of life.
  Total length of CPAP/NIPPV support assessed retrospectively using video recordings (min)
Clinical: Total time on noninvasive and invasive respiratory support | Until 36 weeks postmenstrual age
  Total time on invasive and noninvasive respiratory support (days)
Clinical: Frequency and duration of facemask repositioning | During the first 30 minutes after birth.
  Frequency and duration of facemask repositioning assessed retrospectively using video recordings.
Clinical: Intubation | At 24 and 72 hours of life, at 7 days of life. Until 36 weeks postmenstrual age.
  Intubation rate (%)
Clinical: Time to first intubation | From birth until 36 weeks postmenstrual age.
  Time to first intubation (days, minutes)
Clinical: Number of episodes of desaturation and bradycardia | During the first 24 hours of life.
  Number of episodes of desaturation (SpO2 <80%) and bradycardia (<80 beats per minute)
Clinical: Bronchopulmonary dysplasia (BPD) | At 36 weeks postmenstrual age.
  BPD, maximum grade [number of cases]
Clinical: Intraventricular haemorrhage (IVH) | At 36 weeks postmenstrual age.
  IVH, maximum grade [number of cases]
Clinical: Retinopathy of prematurity (ROP) | At 36 weeks postmenstrual age.
  ROP, maximum grade [number of cases]
Clinical: Necrotizing enterocolitis (NEC) | At 36 weeks postmenstrual age.
  NEC, surgically treated [number of cases]
Clinical: Blood-culture positive sepsis | At 36 weeks postmenstrual age.
  Blood-culture positive sepsis [number of cases]

OTHER OUTCOMES:
Safety: Death | Until 36 weeks postmenstrual age.
  Death [number of cases]
Safety: Pulmonary haemorrhage | Until 36 weeks postmenstrual age.
  Pulmonary haemorrhage [number of cases]
Safety: Air leak | Until 36 weeks postmenstrual age.
  Air leak [number of cases]

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minocchieri S, Berry CA, Pillow JJ; CureNeb Study Team. Nebulised surfactant to reduce severity of respiratory distress: a blinded, parallel, randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2019 May;104(3):F313-F319. doi: 10.1136/archdischild-2018-315051. Epub 2018 Jul 26. PMID 30049729
- [Derived] Gaertner VD, Buchler VL, Waldmann A, Bassler D, Ruegger CM. Deciphering Mechanisms of Respiratory Fetal-to-Neonatal Transition in Very Preterm Infants. Am J Respir Crit Care Med. 2024 Mar 15;209(6):738-747. doi: 10.1164/rccm.202306-1021OC. PMID 38032260
- [Derived] Gaertner VD, Minocchieri S, Waldmann AD, Muhlbacher T, Bassler D, Ruegger CM; SUNSET study group. Prophylactic surfactant nebulisation for the early aeration of the preterm lung: a randomised clinical trial. Arch Dis Child Fetal Neonatal Ed. 2023 May;108(3):217-223. doi: 10.1136/archdischild-2022-324519. Epub 2022 Nov 24. PMID 36424125
- [Derived] Gaertner VD, Waldmann AD, Bassler D, Hooper SB, Ruegger CM. Intrapulmonary Volume Changes during Hiccups versus Spontaneous Breaths in a Preterm Infant. Neonatology. 2022;119(4):525-529. doi: 10.1159/000524194. Epub 2022 Apr 8. PMID 35398844